CLINICAL TRIAL: NCT02327013
Title: Interventional, Randomised, Double-blind, Placebo-controlled, Fixed-dose Study of Vortioxetine in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Investigating the Effect of Vortioxetine in Adult ADHD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15996A
Record Dates: First submitted 2014-12-18; First posted 2014-12-30 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Vortioxetine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- vortioxetine 10 mg tablet (Experimental): In Stage 1, patients will receive vortioxetine 10mg/day for 6 weeks.
  In Stage 2, patients who received vortioxetine 10mg/day in Stage 1 will continue on the same treatment for additionally 6 weeks. Placebo non-responders will be re-randomized to placebo, or vortioxetine 10 or 20mg/day for additionally 6 weeks.
  Interventions: Drug: vortioxetine 10 mg tablet
- vortioxetine 20 mg tablet (Experimental): In Stage 1, patients will receive vortioxetine 20mg/day for 6 weeks.
  In Stage 2, patients who received vortioxetine 20mg/day in Stage 1 will continue on the same treatment for additionally 6 weeks. Placebo non-responders will be re-randomized to placebo, or vortioxetine 10 or 20mg/day for additionally 6 weeks.
  Interventions: Drug: vortioxetine 20 mg tablet
- Placebo tablet (Placebo Comparator): In Stage 1, the patients will receive placebo for 6 weeks.
  In Stage 2, placebo responders will continue on placebo for additionally 6 weeks. Placebo non-responders will be re-randomized to placebo, or vortioxetine 10 or 20mg/day for additionally 6 weeks.
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Drug: vortioxetine 10 mg tablet — Oral tablets, once daily
  Other Names: Brintellix®; Lu AA21004; Trintellix®
  Arms: vortioxetine 10 mg tablet
Drug: vortioxetine 20 mg tablet — Oral tablets, once daily
  Other Names: Brintellix®; Lu AA21004; Trintellix®
  Arms: vortioxetine 20 mg tablet
Other: Placebo tablet — Oral tablets, once daily
  Arms: Placebo tablet

SUMMARY:
The purpose is to determine the effect of vortioxetine treatment on ADHD symptoms in adult patients with ADHD in a 12 weeks study.

DETAILED DESCRIPTION:
The study employed the Sequential Parallel Comparison Design (SPCD), a clinical study design which intend to increase signal detection by using two stages of treatment:

* Stage 1 - first 6 weeks of the 12-weeks treatment period (Visit 2/Baseline 1 to Visit 5/Week 6)
* Stage 2 - last 6 weeks of the 12-weeks treatment period (Visit 5/Baseline 2 to Visit 8/Week 12)

In Stage 1, patients were randomized to placebo or vortioxetine 10 or 20mg. Patients on vortioxetine 10 or 20mg/day during Stage 1 remained on the same treatment in Stage 2. Responders to placebo in Stage 1 remained on Placebo in Stage 2. Patients who were placebo non-responders during Stage 1, defined as patients with a <30% reduction in AISRS total score from Baseline 1, were re-randomized to placebo or vortioxetine 10 or 20mg/day in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing and able to attend study appointments within the specified time windows.
* The patient is an outpatient.
* The patient is diagnosed with a primary diagnosis of ADHD according to the DSM-5™ classification.
* The patient has an AISRS total score ≥24.
* The patient has a CGI-S rating ≥4 (moderately ill or worse).

Exclusion Criteria:

* The patient has previously been treated with vortioxetine.
* The patient has any current psychiatric disorder (DSM-IV-TR™ criteria), other than ADHD, as assessed using the Mini International Neuropsychiatric Interview (MINI).
* The patient has a known first-degree relative with bipolar disorder.
* The patient suffers from intellectual disability as evaluated by the Wechsler Abbreviated Scale of Intelligence (WASI) II vocabulary and matrix.
* The patient suffers from organic mental disorders, or mental disorders due to a general medical condition (DSM-5™ criteria).
* The patient has reported current use of, or has tested positive for, drugs of abuse (opiates, methadone, cocaine, amphetamines [including ecstasy], barbiturates, benzodiazepines, and cannabinoids). If a patient tests positive for opiates due to incidental use of codeine containing medication, as assessed in a clinical interview, the drug screen may be repeated up to three weeks later but the retest result must be available from the central laboratory latest at Visit 2 and has to be negative for this patient to be eligible for enrolment. If a patient tests positive for amphetamines due to his/her ADHD current treatment, as confirmed by a clinical interview, the patient is eligible for enrolment provided this treatment is discontinued two weeks prior to the Baseline Visit.
* The patient has a history of two prior failed (<50% improvement in symptoms) adequate trials of ADHD treatment.
* The patient has any other disorder for which the treatment takes priority over treatment of ADHD or is likely to interfere with study treatment or impair treatment compliance.
* The patient has a history of moderate or severe head trauma or other neurological disorders or systemic medical diseases that are, in the investigator's opinion, likely to affect central nervous system functioning.
* The patient has attempted suicide within the last 6 months or is at significant risk of suicide (either in the opinion of the Investigator or defined as a "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behaviour on the Columbia-Suicide Rating Scale (C-SSRS) within the last 12 months).

Other protocol defined inclusion and exclusion criteria do apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 227 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (15):
- United States (15):
  - US015, Beverly Hills, California
  - US002, Garden Grove, California
  - US004, National City, California
  - US013, Bradenton, Florida
  - US006, Gainesville, Florida
  - US010, Alpharetta, Georgia
  - US014, Libertyville, Illinois
  - US011, Baltimore, Maryland
  - US009, Boston, Massachusetts
  - US016, Las Vegas, Nevada
  - US005, New York, New York
  - US008, New York, New York
  - US001, Austin, Texas
  - US007, Herndon, Virginia
  - US003, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Vortioxetine 10mg: Patients randomized to treatment with vortioxetine 10mg/day in Stage 1 and continued on the same treatment in Stage 2.
- Vortioxetine 20mg: Patients randomized to treatment with vortioxetine 20mg/day in Stage 1 and continued on the same treatment in Stage 2.
- Placebo - Placebo: Patients randomized to treatment with placebo in Stage 1 and continued on the same treatment in Stage 2. This group will consist of placebo responders and placebo non-responders who were re-randomized to Placebo in Stage 2.
- Placebo - Vortioxetine 10mg: Patients that did not respond to placebo in Stage 1 and were re-randomized to treatment with vortioxetine 10mg/day in Stage 2.
- Placebo - Vortioxetine 20mg: Patients that did not respond to placebo in Stage 1 and were re-randomized to treatment with vortioxetine 20mg/day in Stage 2.
Period: Overall Study
Arm/Group | Vortioxetine 10mg | Vortioxetine 20mg | Placebo - Placebo | Placebo - Vortioxetine 10mg | Placebo - Vortioxetine 20mg
Started | 49 | 45 | 96 | 21 | 16
Completed | 36 | 29 | 54 | 20 | 12
Not Completed | 13 | 16 | 42 | 1 | 4
Not completed — Adverse Event | 4 | 4 | 3 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 5 | 0 | 1
Not completed — Non-compliance with IMP | 1 | 2 | 7 | 0 | 0
Not completed — Withdrawal of Consent | 1 | 0 | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 4 | 5 | 0 | 0
Not completed — Administrative or other reason(s) | 1 | 5 | 11 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 3 | 0 | 1
Not completed — Withdrawal before treatment | 2 | 1 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo (Stage 1): Patients treated wtih placebo in Stage 1.
- Vortioxetine 10mg (Stage 1): Patients treated with vortioxetine 10mg in Stage 1.
- Vortioxetine 20mg (Stage 1): Patients treated with vortioxetine 20mg in Stage 1.
- Total: Total of all reporting groups
Arm/Group | Placebo (Stage 1) | Vortioxetine 10mg (Stage 1) | Vortioxetine 20mg (Stage 1) | Total
Number analyzed (Participants) | 128 | 47 | 44 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.3) | 35.8 (9.6) | 37.2 (10.4) | 36.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 24 | 19 | 109
  Male | 62 | 23 | 25 | 110
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 4 | 1 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 15 | 3 | 8 | 26
  White | 97 | 37 | 31 | 165
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in ADHD Investigator Symptom Rating Scale (AISRS) Total Score
Description: AISRS: an 18-item scale administered by the investigator. It included 9 items that evaluated symptoms of inattention and 9 items that evaluated symptoms of impulsivity and hyperactivity. Each item was rated from 0 (none) to 3 (severe). AISRS total score was calculated as sum of all the items on the scale and ranged from 0 to 54. A higher score corresponded to a worse severity of ADHD.
Time Frame: Baseline to Week 6
Population: Stage 2 dataset includes placebo non-responders from Stage 1 that were re-randomized and treated in Stage 2. The statistical analyses were performed on each stage separately, and the combined analysis was performed by constructing a simple equally weighed least square test-statistic.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo, Stage 1: Patients treated with placebo in Stage 1.
- Vortioxetine 10mg, Stage 1: Patients treated with vortioxetine 10mg in Stage 1.
- Vortioxetine 20mg, Stage 1: Patients treated with vortioxetine 20mg in Stage 1.
- Placebo, Stage 2: Placebo responders from Stage 1 continue on placebo in Stage 2.
- Vortioxetine 10mg, Stage 2: Placebo non-responders from Stage 1 re-randomized to treatment with vortioxetine 10mg in Stage 2.
- Vortioxetine 20mg, Stage 2: Placebo non-responders from Stage 1 re-randomized to treatment with vortioxetine 20mg in Stage 2.
- Placebo, Combined: Combined data from patients treated with placebo in Stage 1 and 2
- Vortioxetine 10mg, Combined: Combined data from patients treated with vortioxetine 10mg in Stage 1 and 2
- Vortioxetine 20mg, Combined: Combined data from patients treated with vortioxetine 20mg in Stage 1 and 2
Arm/Group | Placebo, Stage 1 | Vortioxetine 10mg, Stage 1 | Vortioxetine 20mg, Stage 1 | Placebo, Stage 2 | Vortioxetine 10mg, Stage 2 | Vortioxetine 20mg, Stage 2 | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 109 | 41 | 34 | 20 | 20 | 12 | 129 | 61 | 46
units on a scale | -12.4 (1.25) | -12.8 (1.99) | -11.6 (2.17) | -4.1 (1.92) | -3.9 (1.98) | -2.9 (2.35) | -8.3 (1.1) | -8.3 (1.4) | -7.3 (1.6)
Statistical Analysis 1: Comparison: Placebo, Combined vs Vortioxetine 10mg, Combined; The mean difference between treatment groups was estimated based on LS means for the treatment-by-visit interaction in stagewise MMRM analyses. In each stage, the REML-based MMRM model included site ID (stage 1 only), visit, treatment (placebo, vortioxetine 10mg, vortioxetine 20mg), baseline (for the stage) AISRS total score, treatment-by-visit interaction, and baseline (stage) AISRS total score-by-visit interaction, with an unstructured covariance structure to model the within-patient errors; Test type: Superiority; p = 0.9723, weighed z-score; Equally weighed LS z-score, combining results from stagewise MMRM, was compared to standard normal distribution; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-3.6 to 3.5], Standard Error of Mean 1.8
Statistical Analysis 2: Comparison: Placebo, Combined vs Vortioxetine 20mg, Combined; Test type: Superiority — The mean difference between treatment groups was estimated based on LS means for the treatment-by-visit interaction in stagewise MMRM analyses. In each stage, the REML-based MMRM model included site ID (stage 1 only), visit, treatment (placebo, vortioxetine 10mg, vortioxetine 20mg), baseline (for the stage) AISRS total score, treatment-by-visit interaction, and baseline (stage) AISRS total score-by-visit interaction, with an unstructured covariance structure to model the within-patient errors; p = 0.6010, weighed z-score; Equally weighed LS z-score, combining results from stagewise MMRM, was compared to standard normal distribution; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-2.8 to 4.8], Standard Deviation 1.9

2. Secondary Outcome: Inattention/Meta-cognition: Change in Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) Using Metacognition Index
Description: The Metacognition Index (MI) is an index score of the BRIEF-A consisting of 5 scales: initiate, working memory, plan/organise, task monitor, and organization of materials. Each item is rated on a 3-point scale with the numeric score of 1 to 3. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Stage 1 | Vortioxetine 10mg, Stage 1 | Vortioxetine 20mg, Stage 1 | Placebo, Stage 2 | Vortioxetine 10mg, Stage 2 | Vortioxetine 20mg, Stage 2 | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 107 | 41 | 34 | 20 | 20 | 12 | 127 | 61 | 46
T-score | -10.0 (1.26) | -11.2 (1.98) | -10.2 (2.16) | -3.1 (2.28) | -2.6 (2.34) | 0.9 (2.84) | -6.5 (1.3) | -6.9 (1.5) | -4.6 (1.8)

3. Secondary Outcome: Cognitive Function/Global Executive Function: Change in BRIEF-A Using the Global Executive Composite Score
Description: BRIEF-A is a validated questionnaire composed of 75-item within nine non-overlapping scales: 4 scales in the Behavioral Regulation Index (BRI) (inhibit, shift, emotional control, and self-monitor), and 5 scales in the Metacognition Index (MI) (initiate, working memory, plan/organise, task monitor, and organization of materials). Each item is rated on a 3-point scale with the numeric score of 1 to 3. The BRIEF-A yields an overall score (Global Executive Composite) composed of two index scores, the MI and the BRI. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Stage 1 | Vortioxetine 10mg, Stage 1 | Vortioxetine 20mg, Stage 1 | Placebo, Stage 2 | Vortioxetine 10mg, Stage 2 | Vortioxetine 20mg, Stage 2 | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 107 | 41 | 34 | 20 | 20 | 12 | 127 | 61 | 46
T-score | -9.9 (1.22) | -12.5 (1.93) | -11.4 (2.10) | -3.0 (2.24) | -3.5 (2.31) | 2.1 (2.80) | -6.5 (1.3) | -8.0 (1.5) | -4.6 (1.8)

4. Secondary Outcome: Overall Functioning: Change in Sheehan Disability Scale (SDS) Total Score
Description: The SDS comprises a series of patient rated scales designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and 3) home life or family responsibilities are impaired on a 10-point visual analogue scale, on which 0 = normal functioning and 10 = severe functional impairment. The number of days lost and the number of underproductive days last from work/school due to symptoms are also captured. The total score is calculated as a sum of the 3 visual analogue scales, ranges from 0 to 30. A higher score represents more severe functional impairment. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Stage 1 | Vortioxetine 10mg, Stage 1 | Vortioxetine 20mg, Stage 1 | Placebo, Stage 2 | Vortioxetine 10mg, Stage 2 | Vortioxetine 20mg, Stage 2 | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 92 | 34 | 28 | 18 | 17 | 11 | 110 | 51 | 39
units on a scale | -5.3 (0.74) | -7.9 (1.20) | -7.4 (1.29) | 0.6 (0.91) | -0.9 (0.95) | -1.4 (1.14) | -2.4 (0.6) | -4.4 (0.8) | -4.4 (0.9)

5. Secondary Outcome: Productivity: Change in Work Limitations Questionnaire (WLQ) Productivity Loss Score
Description: The WLQ is a patient self-rated scale designed to assess on-the-job impact of chronic health problems and/or treatment. The WLQ consists of 25 items in 4 dimensions: limitations handling time (5 items), physical work demands (6 items), mental-interpersonal work demands (9 items), and output demands (5 items). Each item is rated on a 5-point scale from "All of the Time" (score 5) to "None of the Time" (score 0), or "Does Not Apply to My Job". The WLQ Productivity Loss Score is derived from the Global Productivity Index, which is calculated as a weighed sum of the 4 dimensions. Reduction in WLQ Productivity Loss score indicates less work limitation and represents the estimated percentage of productivity loss in the past two weeks due to presenteeism relative to a healthy benchmark sample. WLQ Productivity Loss Score ranges from 0% to 24,9%.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days lost
Arm/Group | Placebo, Stage 1 | Vortioxetine 10mg, Stage 1 | Vortioxetine 20mg, Stage 1 | Placebo, Stage 2 | Vortioxetine 10mg, Stage 2 | Vortioxetine 20mg, Stage 2 | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 91 | 36 | 27 | 15 | 17 | 11 | 106 | 53 | 38
percentage of days lost | -2.4 (0.54) | -2.5 (0.84) | -2.4 (0.96) | -0.8 (1.02) | -0.9 (0.97) | -0.7 (1.20) | -1.6 (0.6) | -1.7 (0.6) | -1.5 (0.8)

6. Secondary Outcome: Change in AISRS Inattention Sub-score
Description: The AISRS inattentive subscale score consists of 9 items from the AISRS which address inattention. Each item is rated from 0 to 3. The AISRS inattentive subscale score can range from 0 to 27. A higher score corresponds to a worse severity of ADHD inattentiveness.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Stage 1 | Vortioxetine 10mg, Stage 1 | Vortioxetine 20mg, Stage 1 | Placebo, Stage 2 | Vortioxetine 10mg, Stage 2 | Vortioxetine 20mg, Stage 2 | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 109 | 41 | 34 | 20 | 20 | 12 | 129 | 61 | 46
units on a scale | -6.5 (0.71) | -6.0 (1.14) | -5.9 (1.24) | -1.9 (1.2) | -2.0 (1.21) | -1.6 (1.48) | -4.2 (0.7) | -4.0 (0.8) | -3.8 (1.0)

7. Secondary Outcome: Change AISRS Hyperactivity/Impulsivity Sub-score
Description: The AISRS hyperactive/impulsive subscale score consists of 9 items from the AISRS which address hyperactivity and impulsivity. Each item is rated from 0 to 3. The AISRS hyperactive/impulsive subscale score can range from 0 to 27. A higher score corresponds to a worse severity of ADHD hyperactivity/impulsivity.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Stage 1 | Vortioxetine 10mg, Stage 1 | Vortioxetine 20mg, Stage 1 | Placebo, Stage 2 | Vortioxetine 10mg, Stage 2 | Vortioxetine 20mg, Stage 2 | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 109 | 41 | 34 | 20 | 20 | 12 | 129 | 61 | 46
units on a scale | -5.9 (0.62) | -7.0 (0.99) | -5.7 (1.08) | -2.1 (0.93) | -2.0 (0.97) | -1.2 (1.15) | -4.0 (0.6) | -4.5 (0.7) | -3.4 (0.8)

8. Secondary Outcome: Percentage of Patients Responding (Response Defined as 30% or Greater Reduction From Baseline in AISRS Total Score)
Description: as for outcome 1
Time Frame: Baseline to Week 6
Population: Stage 2 dataset includes placebo non-responders from Stage 1 that were re-randomized and treated in Stage 2. The statistical analyses were performed on each stage separately, and the combined response rate was obtained by constructing an equally weighed estimate of the rate combining the two stages.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 145 | 66 | 56
percentage of participants | 30.9 | 27.5 | 23.1

9. Secondary Outcome: Change in Adult ADHD Self-Report Scale (ASRS) Total Score
Description: The Adult ADHD Self-Report Scale (ASRS) is a patient-rated scale designed to assess the ADHD symptoms in adults based on the diagnostic criteria of DSM-IVTM. The ASRS consist of 18 items, each rated on a 5-point scale from "Never" to "Very Often". The categories "Never" and "Rarely" were combined when calculating the total score to mirror the scoring of the AISRS, with 0 representing "Never"/"Rarely" and 3 representing "Very Often". The Total Score ranges from 0 to 54. A reduction in score indicates less severity of ADHD.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | -4.9 (1.0) | -6.5 (1.3) | -3.4 (1.4)

10. Secondary Outcome: Change in Clinical Global Impression - Severity of Illness (CGI-S) Score
Description: The Clinical Global Impression - Severity of Illness (CGI-S) provides the clinician's impression of the patient's current state of mental illness. The clinician uses his or her clinical experience of this patient population to rate the severity of the patient's current mental illness on a 7-point scale ranging from 1 (Normal - not at all ill) to 7 (among the most extremely ill patients). Higher scores indicate worsening.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 129 | 61 | 46
units on a scale | -0.5 (0.1) | -0.7 (0.1) | -0.6 (0.1)

11. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I) Score
Description: The Clinical Global Impression - Global Improvement (CGI-I) provides the clinician's impression of the patient's improvement (or worsening). The clinician assesses the patient's condition relative to a baseline on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Higher scores indicate worsening.
Time Frame: Week 6
Population: CGI-I refers to study baseline and was for this reason analyzed for Stage 1 only.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo, Stage 1: Data from patients treated with placebo in Stage
- Vortioxetine 10mg, Stage 1: Data from patients treated with vortioxetine 10mg in Stage 1
- Vortioxetine 20mg, Stage 1: Data from patients treated with vortioxetine 20mg in Stage 1
Arm/Group | Placebo, Stage 1 | Vortioxetine 10mg, Stage 1 | Vortioxetine 20mg, Stage 1
Number analyzed (Participants) | 124 | 46 | 40
units on a scale | 3.01 (0.11) | 2.93 (0.17) | 3.15 (0.18)

12. Secondary Outcome: Response (Defined as a CGI-I Score of 1 or 2), Stage 1
Description: as for outcome 11
Time Frame: Week 6
Population: CGI-I refers to study baseline and was for this reason analyzed for Stage 1 only.
Measure: Number; unit: percentages of participants
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 124 | 46 | 40
percentages of participants | 43 | 13 | 11

13. Secondary Outcome: Change in BRIEF-A Using the Behavioural Regulation Index
Description: The Behavioral Regulation Index (BRI) is an index score of the BRIEF-A and consists of 4 scales: inhibit, shift, emotional control, and self-monitor). Each item is rated on a 3-point scale with the numeric score of 1 to 3. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
T-score | -5.3 (1.1) | -7.9 (1.3) | -3.9 (1.6)

14. Secondary Outcome: Change in BRIEF-A Subscales - Inhibit
Description: The BRIEF-A subscale Inhibit is a subscale within the Behavioural Regulation Index (BRI). Each item is rated on a 3-point scale ranging from 1 (never) to 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 43
T-score | -5.5 (1.4) | -8.6 (1.5) | -3.2 (1.8)

15. Secondary Outcome: Change BRIEF-A Subscales - Initiate
Description: The BRIEF-A subscale Initiate is a subscale within the Behavioural Regulation Index (BRI). Each item is rated on a 3-point scale ranging from 1 (never) to 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
T-score | -6.2 (1.4) | -5.8 (1.6) | -4.2 (1.8)

16. Secondary Outcome: Change in BRIEF-A Subscales - Organization of Materials
Description: The BRIEF-A subscale Organization of Materials is a subscale within the Behavioural Regulation Index (BRI). Each item is rated on a 3-point scale ranging from 1 (never) to 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
T-score | -4.4 (1.1) | -6.3 (1.3) | -3.2 (1.5)

17. Secondary Outcome: Change in BRIEF-A Subscales - Planning/Organize
Description: The BRIEF-A subscale Planning/Organize is a subscale within the Behavioural Regulation Index (BRI). Each item is rated on a 3-point scale ranging from 1 (never) to 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
T-score | -8.2 (1.6) | -8.7 (1.8) | -6.8 (2.1)

18. Secondary Outcome: Change in BRIEF-A Subscales - Shift
Description: The BRIEF-A subscale Shift is a subscale within the Behavioural Regulation Index (BRI). Each item is rated on a 3-point scale ranging from 1 (never) to 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
T-score | -5.6 (1.4) | -9.1 (1.6) | -3.5 (1.9)

19. Secondary Outcome: Change in BRIEF-A Subscales - Self Monitor
Description: The BRIEF-A subscale Self Monitor is a subscale within the Behavioural Regulation Index (BRI). Each item is rated on a 3-point scale ranging from 1 (never) to 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
T-score | -6.5 (1.4) | -11.0 (1.6) | -4.8 (1.8)

20. Secondary Outcome: Change in BRIEF-A Subscales - Task Monitor
Description: The BRIEF-A subscale Task Monitor is a subscale within the Behavioural Regulation Index (BRI). Each item is rated on a 3-point scale ranging from 1 (never) to 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
T-score | -6.4 (1.5) | -7.8 (1.7) | -4.9 (2.0)

21. Secondary Outcome: Change in BRIEF-A Subscales - Working Memory
Description: The BRIEF-A subscale Working Memory is a subscale within the Behavioural Regulation Index (BRI). Each item is rated on a 3-point scale ranging from 1 (never) to 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
T-score | -7.6 (1.6) | -9.9 (1.8) | -3.8 (2.1)

22. Secondary Outcome: Change in BRIEF-A Subscales - Emotional Control
Description: The BRIEF-A subscale Emotional Control is a subscale within the Behavioural Regulation Index (BRI). Each item is rated on a 3-point scale ranging from 1 (never) to 3 (often). Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
T-score | -3.4 (1.0) | -4.8 (1.1) | -3.5 (1.4)

23. Secondary Outcome: Change in Perceived Deficits Questionnaire - Depression (PDQ-D) Total Score
Description: The PDQ-D is a patient-rated scale designed to assess cognitive impairment/dysfunction adapted for MDD. Each item is rated on a scale from 0 (never) to 4 (almost always). The total score of the 20 items ranges from 0 to 80 with higher scores reflect greater subjective cognitive impairment. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | -7.6 (1.6) | -9.3 (2.0) | -6.3 (2.2)

24. Secondary Outcome: Change in PDQ-D Subscales - Attention and Concentration Sub-score
Description: The PDQ-D attention/concentration sub-score consists of items 1, 5, 9, 13, and 17 of the PDQ with a score ranging from 0 to 20. A higher score reflects greater subjective cognitive impairment. A reduction in score indicates less cognitive impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | -1.7 (0.4) | -2.3 (0.5) | -1.8 (0.6)

25. Secondary Outcome: Change in PDQ-D Sub-scales - Retrospective Memory Sub-score
Description: The PDQ-D retrospective memory sub-score consists of items 2, 6, 10, 14, and 18 of the PDQ (see Outcome 23) with a score ranging from 0 to 20. A higher score reflects greater subjective cognitive impairment. A reduction in score indicates less cognitive impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | -1.8 (0.5) | -2.4 (0.6) | -1.5 (0.6)

26. Secondary Outcome: Change in PDQ-D Sub-scales - Prospective Memory Sub-score
Description: The PDQ-D prospective memory sub-score consists of items 3, 7, 11, 15, and 19 of the PDQ (see Outcome 23) with a score ranging from 0 to 20. A higher score reflects greater subjective cognitive impairment. A reduction in score indicates less cognitive impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | -1.5 (0.4) | -2.3 (0.5) | -0.9 (0.6)

27. Secondary Outcome: Change in PDQ-D Sub-scales - Planning and Organisation Sub-score
Description: The PDQ-D planning and organisation sub-score consists of items 4, 8, 12, 16, and 20 of the PDQ (see Outcome 23) with a score ranging from 0 to 20. A higher score reflects greater subjective cognitive impairment. A reduction in score indicates less cognitive impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | -2.4 (0.5) | -2.5 (0.6) | -1.9 (0.7)

28. Secondary Outcome: Change in SDS Item Scores - Family
Description: The SDS item family is rated from 0 = normal functioning to 10 = severe functional impairment (see outcome 4). A higher score represents more severe functional impairment. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
units on a scale | -1.5 (0.3) | -1.8 (0.3) | -1.5 (0.4)

29. Secondary Outcome: Change in SDS Item Scores - Work
Description: The SDS item work is rated from 0 = normal functioning to 10 = severe functional impairment (see outcome 4). A higher score represents more severe functional impairment. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 109 | 50 | 38
units on a scale | -1.2 (0.3) | -2.0 (0.4) | -2.1 (0.4)

30. Secondary Outcome: Change in SDS Item Scores - Social Life
Description: The SDS item social life is rated from 0 = normal functioning to 10 = severe functional impairment (see outcome 4). A higher score represents more severe functional impairment. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
units on a scale | -1.1 (0.3) | -1.7 (0.3) | -1.5 (0.4)

31. Secondary Outcome: Change in SDS Item Scores - Number of Days Lost
Description: This SDS item captures days lost from school or work (see outcome 4).
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
days | -0.3 (0.1) | -0.2 (0.1) | -0.1 (0.2)

32. Secondary Outcome: Change in SDS Item Scores - Number of Underproductive Days
Description: This SDS item captures the number of underproductive days (see outcome 4)
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 127 | 61 | 46
days | -1.2 (0.3) | -1.0 (0.3) | -1.2 (0.3)

33. Secondary Outcome: Change in WLQ Using the Global Productivity Index
Description: The WLQ is a patient self-rated scale designed to assess on-the-job impact of chronic health problems and/or treatment. The WLQ consists of 25 items in 4 dimensions: limitations handling time (5 items), physical work demands (6 items), mental-interpersonal work demands (9 items), and output demands (5 items). Each item is rated on a 5-point scale from "All of the Time" (score 5) to "None of the Time" (score 0), or "Does Not Apply to My Job". The Global Productivity Index is calculated as a weighed sum of the 4 dimensions, and ranges from 0.000 to 0.286. Reduction in score indicates less work limitation.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Index
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 106 | 53 | 37
Index | -0.0 (0.0) | -0.0 (0.0) | -0.0 (0.0)

34. Secondary Outcome: Change in WLQ Domain Scores - Limitations Handling Time
Description: Limitations Handling Time is scored on a scale of 0 (limited at work none of the time) to 100 (limited at work all of the time) based on a converted mean score. A reduction in score indicates less work limitation.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 117 | 57 | 43
units on a scale | -5.6 (2.7) | -7.7 (3.1) | -2.2 (3.7)

35. Secondary Outcome: Change in WLQ Domain Scores - Mental-Interpersonal Work Demands
Description: Mental-Interpersonal Work Demands is scored on a scale of 0 (limited at work none of the time) to 100 (limited at work all of the time) based on a converted mean score. A reduction in score indicates less work limitation.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 126 | 59 | 49
units on a scale | -8.4 (2.2) | -8.2 (2.6) | -6.2 (2.9)

36. Secondary Outcome: Change in WLQ Domain Scores - Physical Demands
Description: Physical Demands is scored on a scale of 0 (limited at work none of the time) to 100 (limited at work all of the time) based on a converted mean score. A reduction in score indicates less work limitation.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 115 | 53 | 43
units on a scale | -5.5 (2.4) | -5.0 (2.9) | -4.6 (3.2)

37. Secondary Outcome: Change in WLQ Domain Scores - Output Demands
Description: Output Demands is scored on a scale of 0 (limited at work none of the time) to 100 (limited at work all of the time) based on a converted mean score. A reduction in score indicates less work limitation.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 122 | 57 | 47
units on a scale | -8.9 (3.1) | -7.1 (3.5) | -7.2 (4.0)

38. Secondary Outcome: Change in Adult ADHD Quality of Life Measure (AAQoL) Total Score
Description: The AAQoL is a patient-rated scale designed to assess health-related quality of life in adults with ADHD. The AAQoL consists of 29 items, each item is rated on a 5-point scale from 1 (not at all/never) to 5 (extremely/very often). The AAQoL Total score is based on all 29 items and ranges from 29 to 145. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | 7.7 (1.7) | 9.1 (2.1) | 5.4 (2.3)

39. Secondary Outcome: Change in AAQoL Subscales - Life Productivity Sub-score
Description: The AAQoL is a patient-rated scale designed to assess health-related quality of life in adults with ADHD. The AAQoL consists of 29 items, each item is rated on a 5-point scale from 1 (not at all/never) to 5 (extremely/very often). The AAQoL Life productivity subscale is based on 11 items and ranges from 11 to 55. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | 10.9 (2.4) | 11.6 (2.8) | 6.4 (3.1)

40. Secondary Outcome: Change in AAQoL Subscales - Psychological Health Sub-score
Description: The AAQoL is a patient-rated scale designed to assess health-related quality of life in adults with ADHD. The AAQoL consists of 29 items, each item is rated on a 5-point scale from 1 (not at all/never) to 5 (extremely/very often). The AAQoL Psychological Health subscale is based on 6 items and ranges from 6 to 30. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | 6.7 (2.2) | 10.3 (2.5) | 5.7 (2.7)

41. Secondary Outcome: Change in AAQoL Subscales - Life Outlook Sub-score
Description: The AAQoL is a patient-rated scale designed to assess health-related quality of life in adults with ADHD. The AAQoL consists of 29 items, each item is rated on a 5-point scale from 1 (not at all/never) to 5 (extremely/very often). The AAQoL Life Outlook subscale is based on 7 items and ranges from 7 to 35. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | 3.7 (1.3) | 5.0 (1.7) | 3.0 (1.8)

42. Secondary Outcome: Change in AAQoL Subscales - Relationships Sub-score
Description: The AAQoL is a patient-rated scale designed to assess health-related quality of life in adults with ADHD. The AAQoL consists of 29 items, each item is rated on a 5-point scale from 1 (not at all/never) to 5 (extremely/very often). The AAQoL Relationship subscale is based on 5 items and ranges from 5 to 25. A reduction in score indicates less impairment.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo, Combined | Vortioxetine 10mg, Combined | Vortioxetine 20mg, Combined
Number analyzed (Participants) | 132 | 62 | 53
units on a scale | 7.4 (2.1) | 8.1 (2.5) | 6.0 (2.7)

ADVERSE EVENTS:
Time Frame: Baseline to end of study (16 weeks)
Description: Treatment-Emergent Adverse Events are reported in this section
Groups:
- Placebo-Placebo: Patients randomized to treatment with placebo in Stage 1 and continued on the same treatment in Stage 2. This group consists of placebo responders and placebo non-responders who were re-randomized to Placebo in Stage 2.
- Vortioxetine 10mg: Patients randomized to treatment with vortioxetine 10mg/day in Stage 1 and continued on the same treatment in Stage 2. In addition, patients that did not respond to placebo in Stage 1 and were re-randomized to treatment with vortioxetine 10mg/day in Stage 2.This group consists of patients who had received dosing of 10 mg vortioxetine in the study.
- Vortioxetine 20mg: Patients randomized to treatment with vortioxetine 20mg/day in Stage 1 and continued on the same treatment in Stage 2. In addition, patients that did not respond to placebo in Stage 1 and were re-randomized to treatment with vortioxetine 20mg/day in Stage 2. This group consists of patients who had received dosing of 20 mg vortioxetine in the study.
Arm/Group | Placebo-Placebo | Vortioxetine 10mg | Vortioxetine 20mg
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/68 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/91 | 1/68 | 0/60
Other Adverse Events (participants affected / at risk) | 39/91 | 34/68 | 36/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Placebo (N=91) | Vortioxetine 10mg (N=68) | Vortioxetine 20mg (N=60)
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Placebo (N=91) | Vortioxetine 10mg (N=68) | Vortioxetine 20mg (N=60)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 5
Nausea (Gastrointestinal disorders) | 3 | 15 | 18
Vomiting (Gastrointestinal disorders) | 1 | 4 | 3
Fatigue (General disorders) | 10 | 7 | 11
Nasopharyngitis (Infections and infestations) | 4 | 2 | 4
Weight increased (Investigations) | 2 | 5 | 3
Dizziness (Nervous system disorders) | 4 | 4 | 2
Headache (Nervous system disorders) | 17 | 10 | 10
Somnolence (Nervous system disorders) | 3 | 1 | 3
Insomnia (Psychiatric disorders) | 9 | 4 | 5

LIMITATIONS AND CAVEATS:
Combined analysis: the overall number of participants analyzed corresponds to the total number of patients in the two stage-wise analyses, where Stage 2 includes patients already included in Stage 1 (patient data not used in the combined analysis).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No